CLINICAL TRIAL: NCT00231270
Title: Stenting and Angioplasty With Protection in Patients at High Risk for Endarterectomy
Brief Title: Stenting and Angioplasty With Protection in Patients at High Risk for Endarterectomy (SAPPHIRE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P98-5201
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2007-07

CONDITIONS: Carotid Artery Disease
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cordis Nitinol Stent
Device: PRECISE tapered stent
Device: ANGIOGUARD XP Emboli Capture Guidewire (ECGW)

SUMMARY:
The primary objective of this study is to compare the safety and effectiveness of the Cordis Nitinol Carotid Stent and Delivery Systems (5.5 F and 7 F) with the ANGIOGUARD XP distal protective device to CEA in the treatment of carotid artery disease in patients at increased risk for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be > 18 years of age.
2. The patient has a 50% stenosis (as determined by ultrasound or angiogram) of the common or internal carotid artery and is clinically symptomatic; i.e., within the previous 180 days has experienced symptoms in the ipsilateral carotid artery distribution, defined as:

   * one or more TIAs, characterized by distinct focal neurologic dysfunction or monocular blindness with clearing of signs and symptoms within 24 hours, or
   * one or more completed strokes (as defined by this protocol) with persistence of symptoms or signs for more than 24 hours (the most recent event is used as the qualifying event), except as excluded below, with stenosis >50%, (as determined by ultrasound or angiogram) of the common or internal carotid artery, OR The patient must have a >80% diameter stenosis (as determined by ultrasound or angiogram) of the internal or common carotid artery without neurological symptoms.
3. To be entered into the study, the patient must have one or more of the following conditions:

   * congestive heart failure (class III/IV) and/or known severe left ventricular dysfunction LVEF < 30%
   * open heart surgery within six weeks
   * recent MI (>24 hours and <4 weeks)
   * unstable angina (CCS class III/IV)
   * synchronous severe cardiac and carotid disease requiring open heart surgery and carotid revascularization
   * Age greater than 80 years as a single risk factor.

Exclusion Criteria:

1. The patient is experiencing an acute ischemic neurologic stroke or has experienced a stroke within the past 48 hours.
2. The patient has an intracranial mass lesion (i.e., abscess, tumor, or infection).
3. The reference segment diameter (distal common carotid and internal carotid artery segment cephalic to the lesion) is less than 4mm or greater than 9mm by quantitative analysis. See Instructions For Use, for proper stent sizing. The exception to this would be with a lesion having >95% stenosis where the true diameter of the distal vessel can not be determined such as the case with a string sign or distal vessel collapse. In this case the judgment of the interventionalist will prevail with the intention not to oversize the stent to the distal vessel by more than 2mm.
4. The patient has known peripheral vascular, supra-aortic or internal carotid artery tortuosity which preclude the use of catheter-based techniques if so randomized.
5. The patient has any intracranial aneurysm (> 9 mm).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300
Dates: Start 2000-08; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
composite of major adverse clinical events including death, any stroke, and/or myocardial infarction at 30-days post-procedure | 30-days post-procedure
The same 30-day composite of major adverse clinical events plus death and/or ipsilateral stroke between 31-days and 12-months post-procedure. | Between day 31 and 12-months post-procedure.

SECONDARY OUTCOMES:
successful stent deployment at the target lesion in a variety of carotid morphologies
successful filter deployment and retrieval
<30% residual stenosis determined by angiography immediately post-stent placement and post-dilatation
endovascular access site complications, such as the need for surgical repair or blood transfusion
surgical site complications, such as wound infection or hematoma, that prolong hospital stay, require incision and drainage, or need blood transfusion
patency (< 50% restenosis) of the Cordis Nitinol Stent as determined by carotid ultrasound imaging within 48 hours, at six months, and one, two and three years post-procedure
independent neurologic assessments at 24 + 12 hours, thirty days, six months, and one, two and three years post-procedure (in addition to stroke scales, the development of any cranial nerve deficits will be recorded) - persistent neurologic deficits
thirty (30)-day and six (6)-month evaluation for disabling stroke | Day 30 and 6 months
six (6)-month, one (1)-year, two (2)-year and three (3)-year composite of major adverse clinical events including death and ipsilateral stroke | 6 month and 1, 2, 3yr
safety assessment of the ANGIOGUARD XP Emboli Capture Guidewire Device
presence of trapped material as determined by the interventionalist's visual inspection of the ANGIOGUARD XP filter basket following recapture at the completion of the procedure
laboratory analysis of trapped material contained in the ANGIOGUARD XP filter basket

REFERENCES:
- [Result] Yadav JS, Wholey MH, Kuntz RE, Fayad P, Katzen BT, Mishkel GJ, Bajwa TK, Whitlow P, Strickman NE, Jaff MR, Popma JJ, Snead DB, Cutlip DE, Firth BG, Ouriel K; Stenting and Angioplasty with Protection in Patients at High Risk for Endarterectomy Investigators. Protected carotid-artery stenting versus endarterectomy in high-risk patients. N Engl J Med. 2004 Oct 7;351(15):1493-501. doi: 10.1056/NEJMoa040127. PMID 15470212
- [Result] Gurm HS, Yadav JS, Fayad P, Katzen BT, Mishkel GJ, Bajwa TK, Ansel G, Strickman NE, Wang H, Cohen SA, Massaro JM, Cutlip DE; SAPPHIRE Investigators. Long-term results of carotid stenting versus endarterectomy in high-risk patients. N Engl J Med. 2008 Apr 10;358(15):1572-9. doi: 10.1056/NEJMoa0708028. PMID 18403765